CLINICAL TRIAL: NCT06178575
Title: Apply Machine Learning to the Interpretation of Urinary Crystal Morphology.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yi-Shiou Tseng (Other)
Responsible Party: Sponsor-Investigator, Yi-Shiou Tseng, Attending physician, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Other Study IDs: 112183-E
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Kidney Calculi
Keywords: machine learning; urinary crystal
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manual microscopic observation: Control Group: Manual analysis of urine crystal images, distinguishing crystal types, recording accuracy, and analyzing the time consumed.
- Machine interpretation: The urine crystal images undergo analysis for crystal types, followed by image preprocessing and category labeling for machine software learning and inference. Subsequently, the interpreted results will be subjected to statistical analysis software to assess accuracy.

SUMMARY:
The goal of this observational study is to developing an image-based artificial intelligence software that can automatically interpret the types and sizes of crystals in urine. The main question[s] it aims to answer are:

* Allowing healthcare professionals to input urine images and receive real-time reading results on crystal types and sizes.
* This aims to provide a faster, more objective, and accurate analysis of crystals.

We anticipate delivering an image AI software suitable for practical applications, promoting the automation and accuracy of urine crystal analysis.

DETAILED DESCRIPTION:
Kidney stones are primarily formed due to the supersaturation of ions in urine, leading to the formation of crystals. An assessment of the risk of kidney stones is based on a patient's medical history, biochemical urine tests, and various laboratory examinations. Combining these with imaging studies such as CT scans, ultrasound, and X-rays helps in diagnosing the type of kidney stones, though imaging results for smaller stones may be less accurate. Stone formation is common with a high recurrence rate, and there is a strong correlation between urine crystals and stone composition. Therefore, the analysis of urine crystals is meaningful for the diagnosis, evaluation of treatment strategies, and prevention of stone recurrence in kidney stone disease.

Microscopic analysis of urine crystals allows the observation of smaller crystals. However, manual urine microscopy is slow and time-consuming. To address this, we aim to develop artificial intelligence software to assist in the interpretation of urine crystals, providing a faster analysis. We will retrospectively analyze urine crystal images stored from previous research (Chang Gung Memorial Hospital Internal Project Research No. 107123-E) to identify crystal types. Subsequent image preprocessing and category labeling will be done to train and infer machine software. The results will be compared with manual interpretation to establish the accuracy of the software.

ELIGIBILITY:
Inclusion Criteria:

* Retrospectively analyze the urine crystal images preserved from the previous study 107123-E for crystal type analysis. Subsequently, conduct image preprocessing and label categorization for machine software learning and inference. The interpreted results will then be assessed for accuracy using statistical analysis software.

Exclusion Criteria:

* Not applicable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Calcium oxalate kidney stone patient
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Kappa statistics | The machine requires approximately 0.5 hours to complete the interpretation of around 800 urine crystal images.
  Used for comparing between a new instrument and a standard instrument to determine whether the new instrument exhibits a certain level of performance or accuracy.

IPD SHARING:
Plan to Share IPD: No
This study involves retrospectively analyzing urine crystal images preserved from a previous study (Intramural Research Project Code 107123-E at Far Eastern Memorial Hospital). Subsequently, image preprocessing and category labeling will be applied to facilitate machine software learning and inference. The interpreted results will then undergo statistical analysis for accuracy using dedicated software. Participant information and experimental data are stored on a computer in a shared laboratory, with access secured through password protection to ensure data security. Participant identities are encoded for confidentiality. Once the required information is collected, the original participant identities will be linked with their respective codes. Researchers will not obtain the list of potential participants through privacy-invasive means.